CLINICAL TRIAL: NCT05815134
Title: Cell Free DNA Quantification in Patients With Endometriosis Followed Witd Medical Assistance to Procreation
Acronym: ENDO-FIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PI2019_843_0087
Record Dates: First submitted 2023-03-20; First posted 2023-04-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Endometriosis; Cell Free DNA
Keywords: Endometriosis; cell free DNA; oocyte quality
MeSH Terms: conditions — Endometriosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with endometriosis (Experimental)
  Interventions: Biological: blood sample
- others infertility causes (Active Comparator)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — 10ml of blood will be sampled from patients before undergoing IVF treatment, the cell free DNA will be extracted and then quantified by a real time PCR. Another 10ml sample will be drawn the day of oocyte puncture for a new quantification of cell free DNA in plasma and cell free DNA will also be dose in follicular fluid of patients

SUMMARY:
Endometriosis is a common benign disease in premenopausal women and causes chronic pelvic pain and infertility. This infertility may be due to pelvic adhesions and surgery but also because of poor oocyte quality. It is known that endometriosis is associated with an increase oxidative stress, wich induce chronic inflammation, deleterious effect for DNA, proteins and can caused cellular death. ROS markers found in follicular fluid or in serum are significatively higher in endometriosis women. The investigators want to dose a marker of apoptosis in infertile women and see if it's significatively higher in serum and in follicular fluid of patients with endometriosis compared to others infertility causes and if it's correlated to oocyte quality and IVF results. Real time PCR will be used to dose cell free DNA in serum and follicular fluid of patients undergoing IVF treatment (endometriosis and infertility due to tubal factor, male infertility or idiopathic cause). Then the investigators will compare cell free DNA rate with oocyte and embryo quality and with pregnancy outcomes in the different group.

ELIGIBILITY:
Inclusion Criteria:

* patients eligible medical assistance to procreation who are about to undergo IVF treatment
* aged between 18 and 43 years old
* and who have signed a consent form

Exclusion Criteria:

* patients who are not eligible for medical assistance to procreation,
* patients who are followed for other inflammatory disease,
* patients followed for premature ovarian failure or
* patients with a recent story of pelvic infection

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 114 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
cell free DNA rate in serum in patients before they start IVF stimulation | day 1
  cell free DNA in serum quantified by real time PCR in patients before they start IVF stimulation
cell free DNA rate in follicular fluid the day of punction | day 1
  cell free DNA in follicular fluid the day of punction

SECONDARY OUTCOMES:
number of oocytes reaching the metaphase II | 1 year
  number of oocytes reaching the metaphase II in both groups of patients
fragmentation rate | 1 year
  fragmentation rate
number of cells at day 2 | day 2
  number of cells at day 2
number of cells at day 3 | day 3
  number of cells at day 3
blastulation rate at day 5 of developement | day 5
  blastulation rate at day 5 of developement
number of clinical pregnancy in both groups | 1 year
number of live birth in both groups | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] https://dumas.ccsd.cnrs.fr/dumas-03767871v1/file/2022AMIEM032_VANDECANDELAERE_Albane.pdf